CLINICAL TRIAL: NCT06266637
Title: Effect of Physiotherapeutic Scoliosis-Specific Exercise on Lower Limb Biomechanics in Adolescents With Idiopathic Scoliosis: A Randomised Controlled Trial
Brief Title: Effect of Scoliosis-Specific Exercise on Lower Limb Biomechanics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Ali Elabd, Lecturer of Orthopedic Physical Therapy, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004999
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Scoliosis Idiopathic
Keywords: scoliosis; exercise; lower limb; biomechanics
MeSH Terms: conditions — Scoliosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The experimental group will receive the same standard treatment in addition to Physiotherapeutic Scoliosis-Specific Exercise
  Interventions: Other: Conventional Physical Therapy Program; Other: Physiotherapeutic Scoliosis-Specific Exercise (Schroth)
- Control group (Active Comparator): The control group will receive the standard care composed of trunk muscles strengthening exercises, trunk proprioception exercises .
  Interventions: Other: Conventional Physical Therapy Program

INTERVENTIONS:
Other: Conventional Physical Therapy Program — Conventional Physical Therapy program:
  trunk muscles strengthening exercises, trunk muscles endurance exercises, trunk proprioception exercises . postural correction exercises. Core exercise Spinal mobility exercises
Other: Physiotherapeutic Scoliosis-Specific Exercise (Schroth) — It uses exercises customized for each patient to return the curved spine to a more natural position. The spine is addressed in all three anatomical planes - sagittal, frontal and transverse. The purpose of the method is to create spinal balance and stability by improving body mechanics and spinal stabilization to prevent further curve progression
  Arms: Study group

SUMMARY:
PURPOSE: To examine the effect of Physiotherapeutic Scoliosis-Specific Exercise on limb biomechanical parameters in adolescents with idiopathic scoliosis. A randomised controlled trial

BACKGROUND:

Adolescent idiopathic scoliosis is one of the most common orthopaedic diseases affecting the spine during adolescence. The efficacy of exercise treatment is controversial. Although evidence suggests that PSSE, which include auto-correction in 3D, integration in daily life, stabilizing the corrected posture, and patient education, could improve some outcomes, effect of PSSE on related biomechanical alterations in lower limbs have not yet been examined.

HYPOTHESES:

Null hypothesis There are no statistically significant effect of Physiotherapeutic Scoliosis-Specific Exercise on lower limb biomechanics in scoliotic adolescents.

RESEARCH QUESTION:

What are the effect of Physiotherapeutic Scoliosis-Specific Exercise on lower limb biomechanics in scoliotic adolescents.?

DETAILED DESCRIPTION:
procedures: A randomized controlled clinical trial will be conducted

Assessment:

x-ray computed scanogram radiography of the whole spine and both lower limbs in standing will be used.

The following measurements will be taken pre and post the treatment program:

For the lumbar spine coronal alignment:

1. Cobb's angle for dorso-lumbar scoliosis (curve apex from D10- L4) will be measured.
2. Coronal balance estimated by the distance between plumb line and central sacral line from anterioposterior x-ray view

For both lower limbs:

1. the length will be measured for the limb, the tibia and the femur
2. tibiofemoral angle
3. joint line convergence angle
4. mechanical axis
5. mechanical axis deviation

Treatment:

Patients will be randomly assigned into two groups to receive the prescribed treatment program for 6 months., 1 session per week in addition to a home program of daily exercise .

The control group will receive the standard care composed of trunk muscles strengthening exercises, trunk proprioception exercises .

The experimental group will receive the same standard treatment in addition to Physiotherapeutic Scoliosis-Specific Exercise

Data will be analyzed using 2 way MANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with age 10-18 years
* complaining of dorsolumbar scoliosis
* curves (apex lies between D10 and L4)
* curve magnitudes greater than 15 degrees and less than 90
* using or not using brace
* all maturity levels (Risser = 0-5)

Exclusion Criteria:

* Other types of scoliosis ; congenital or neuromuscular
* Current physical therapy or medical treatment for scoliosis,
* Contracture or surgery affecting the lumbar spine or lower limbs
* Pathologies such as inflammatory diseases
* congenital anomalies
* Neurological disorders like cerebral palsy or ataxia
* dislocations
* visual or auditory problems

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Cobb's angle | From enrollment to the end of treatment at 6 months
  Cobb's angle for dorso-lumbar scoliosis. The angle of the curve apex from D10 to L4 will be assessed by computed radiograph (X-ray computed scanogram)
Coronal balance | From enrollment to the end of treatment at 6 months
  Coronal balance estimated by the distance between plumb line and central sacral line from Anetroposterior x-ray view assessed by computed radiograph (X-ray computed scanogram )
length of the the tibia and femur | From enrollment to the end of treatment at 6 months
  The length (in centimeter) of the Tibia and femur will be assessed by computed radiograph (X-ray computed scan-gram)
tibiofemoral angle | From enrollment to the end of treatment at 6 months
  The tibiofemoral angle (TFA), or knee angle, is defined as the angle between the anatomical axis of femur with the anatomical axis of tibia. It will be assessed (in degrees) by computed radiograph (X-ray computed scan-gram)
knee joint line convergence angle | From enrollment to the end of treatment at 6 months
  The knee joint-line convergence angle (KJLCA) h is the angle made by a tangential line between the femoral condyles and the tibial plateau. It will be assessed (in degrees) by computed radiograph (X-ray computed scan-gram)
lower limb mechanical axis; and mechanical axis deviation | From enrollment to the end of treatment at 6 months
  The mechanical axis of the lower limb, also called the Mikulicz line, is drawn by connecting a point in the center of the femoral head to a point in the center of the ankle. The value of the deviation is measured in millimeters and is named mechanical axis deviation (MAD). It will be assessed by computed radiograph (X-ray computed scan-gram).

CONTACTS AND LOCATIONS:
Locations (1):
- Delta university for science and technology, Gamasa, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
personal preferences